CLINICAL TRIAL: NCT01925729
Title: Middle Ear Pressure Regulation in Health and Disease -- Gas Supply, Demand and Middle Ear Gas Balance -- Specific Aim 2
Brief Title: TransMEM Gas Exchange -- Project 1, Aim 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cuneyt M. Alper (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Cuneyt M. Alper, Professor of Otolaryngology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRO13040386; 2P50DC007667-07 (NIH)
Record Dates: First submitted 2013-08-08; First posted 2013-08-20 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Middle Ear Disease; Nasal Allergy
Keywords: middle ear; allergy; nose
MeSH Terms: conditions — Hypersensitivity | interventions — Histamine; Pseudoephedrine; Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ragweed (Experimental): ragweed -- 1000PNU intranasal spray
  Interventions: Biological: ragweed
- histamine (Experimental): 5 mg intranasal spray
  Interventions: Biological: histamine
- pseudoephedrine (Experimental): pseudoephedrine -- 60 mg orally
  Interventions: Drug: pseudoephedrine
- oxymetazoline (Experimental): oxymetazoline 0.05% solution intranasal spray
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Biological: ragweed — ragweed arm only
  Arms: ragweed
Biological: histamine — histamine arm only
  Arms: histamine
Drug: pseudoephedrine — pseudoephedrine arm only
  Other Names: Sudafed
  Arms: pseudoephedrine
Drug: Oxymetazoline — oxymetazoline arm only
  Other Names: Afrin
  Arms: oxymetazoline

SUMMARY:
This study will determine if exposure to an allergy material (ragweed) or exposure to an allergic-symptom-provoking substance (histamine) and medications typically used to decongest the nose changes the rate of blood-flow in the lining of the middle-ear. Otitis media (the build-up of water-like fluid in the middle-ear airspace) may occur if the blood flow in the lining of the middle-ear is too high and may be prevented if a way could be found to lower the blood flow in persons susceptible to the disease. Middle-ear blood flow is measured indirectly by measuring the change in middle-ear pressure while a person breathes a gas mixture containing nitrous oxide ("laughing gas"). In this study, 4 groups of subjects will be entered and middle-ear pressure in persons breathing a mixture of 50% Oxygen, 50% Nitrous Oxide ("laughing gas")will be measured after exposure to one of four substances (ragweed, histamine,an oral decongestant, a decongestant nasal spray) and a fake medication (placebo) at separate test sessions. All subjects will have one set of 2 x-rays of the middle ears and mastoids. The group exposed to ragweed will require 3 study visits while the other 3 groups will have 2 study visits. From this information middle-ear blood flow will be calculated. This will help determine the relationship between what happens in the nose and what happens in the middle ear.

DETAILED DESCRIPTION:
The set of four experiments described here is a subcomponent of one Project included in a Clinical Research Center Grant Program focused on the physiology and pathophysiology of middle-ear (ME) pressure-regulation in children and adults. These experiments are designed to measure the rate of transME mucosal (transMEM) inert gas exchange in adults and determine if nasal inflammatory reactions experimentally provoked by intranasal histamine or allergen challenge increase the rate transMEM inert gas exchange and if nasal or oral treatment with an adrenergic agonist decreases that rate. Four cohorts of 20 otherwise healthy adults will be identified and one cohort assigned to each of the four experiments. All subjects will have a x-ray in Schuller projection to estimate mastoid volume. The transMEM inert gas exchange rate is measured by repeatedly recording ME pressure by tympanometry while the subject breathes a mixture of 50%N2O/ 50%O2, and then regressing ME pressure on time and dividing the slope of the function by the estimated N2O driving gradient to yield an exchange constant. For each experiment, the transMEM N2O exchange rate is measured twice at separate visits (active and placebo). The four experimental conditions are: (1) intranasal ragweed and placebo challenges; (2) intranasal histamine and placebo challenges; (3) oral pseudoephedrine and placebo; (4) intranasal oxymetazoline and placebo. Experiments 2-4 require two visits, while Experiment 1 will require an additional visit to obtain blood for RAST testing to verify ragweed allergy. The paired exchange constants measured in each experiment will be compared for a significant difference using a Student's Paired t test and the results interpreted as supporting or refuting the possibility of modulating the transMEM N2O exchange rate by the different procedures.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* no evidence of otitis media at entry
* bilaterally intact tympanic membranes
* ragweed arm: history of symptomatic ragweed allergy and Class 2 positive on RAST testing with or without other allergic sensitivities by history

Exclusion Criteria:

* craniofacial syndrome (ef, cleft palate)
* Use of prescription medications (except for birth control) in the 1 month prior to entry;
* Use of over-the-counter allergy medication within 2 weeks before challenge (Experiments 1, 2 only);
* Use of over-the-counter decongestants (nasal or oral) within 2 weeks before challenge (Exp 3,4 only)
* Elevated blood pressure (>140/90);
* Individuals with any pulmonary or cardiac problems, including asthma;
* Individuals who are pregnant or who are planning to become pregnant during the period of study;
* Individuals who had immunotherapy for ragweed allergy at any time (Experiment 1 only);
* Individuals who used any experimental medication or treatment within 3 months of screening;
* Individuals with extant unilateral or bilateral otitis media as documented by otoscopy or tympanometry;
* Individuals with abnormally low tympanic membrane mobility, eg Type B tympanogram;
* Individuals reporting a previous adverse experience with breathing gas mixtures containing N2O (e.g. during dental procedures);
* Individuals who have upper respiratory ("cold") symptoms or allergic rhinitis symptoms (may be rescheduled);
* Individuals with single or multiple allergic sensitivities by screening history (Experiment 2 only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
change in trans-middle ear N2O exchange constant | Visit 1 and Visit 2 (Visits 2 and 3 for ragweed arm) up to approximately 3 weeks
  The transMEM N2O exchange constant is the primary outcome measure and is calculated as the slope of the line relating middle-ear pressure to time (until an observable active or passive ET opening) divided by the estimated extant N2O gradient.

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Middle Ear Physiology Laboratory, University of PIttsburgh, Pittsburgh, Pennsylvania, United States